CLINICAL TRIAL: NCT04572997
Title: A Multicenter, Open Label, Single-arm Pilot Study to Evaluate the Efficacy and Safety of Oral Apremilast in Patients With Moderate to Severe Palmoplantar Pustulosis (PPP) (APLANTUS)
Brief Title: Apremilast in Patients With Moderate to Severe Palmoplantar Pustulosis (PPP) (APLANTUS)
Acronym: APLANTUS
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Kristian Reich (Other)
Responsible Party: Sponsor-Investigator, Kristian Reich, Professor Doctor (Prof. Dr.), Universitätsklinikum Hamburg-Eppendorf
Organization: Universitätsklinikum Hamburg-Eppendorf (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 069-008.; 2016-005122-11 (EudraCT Number)
Record Dates: First submitted 2020-09-21; First posted 2020-10-05 (Actual); Results first posted 2021-09-24 (Actual); Last update posted 2021-09-24 (Actual); Status verified 2021-09

CONDITIONS: Palmoplantar Pustulosis
Keywords: PPP; Palmoplantar Pustulosis; Apremilast; Otezla
MeSH Terms: conditions — Psoriasis | interventions — apremilast

STUDY DESIGN:
Intervention Model Description: This was an open-label, single-arm, pilot study to evaluate the efficacy and safety of apremilast.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Full analysis set (FAS) (Experimental): The full analysis set (FAS) consisted of all patients who received at least one dose of study drug.
  Interventions: Drug: Apremilast

INTERVENTIONS:
Drug: Apremilast — Apremilast was taken orally twice daily (except Day 1). Patients received tablets in blister/bottles sufficient for one month. To mitigate potential gastrointestinal side effects (primarily mild-to-moderate nausea and diarrhoea), dose titration was implemented in this study in accordance with the Summary of Product Characteristics (SmPC). A titration pack included tablets of 10, 20 and 30 mg for a period of one month. During the first 5 days, the dosage was up-titrated. The initial dose on day 1 was 10 mg in the morning; this was increased to 10 mg in the morning and evening on day 2. The evening dose was further increased by 10 mg (to 20 mg) on day 3. On day 4, the morning dose was increased to 20 mg, so that 20 mg was taken twice daily, and on day 5 the evening dose was increased to 30 mg. From Day 6 onwards, patients received the 30 mg dose twice a day. Subsequent packs included only tablets of 30 mg strength.
  Other Names: Otezla®

SUMMARY:
Multicenter, open-label, single-arm, phase II, pilot study. The screening period was up to 4 weeks and treatment took place over 20 weeks per patient. Five visits per patient were performed including: Visit 1 at week -4 to -1 (screening), Visit 2 at week 0 (baseline), Visit 3 at week 4, Visit 4 at week 12, and Visit 5 at week 20 (end of study). There was no follow-up period.

DETAILED DESCRIPTION:
This was a multicenter, open-label, single-arm, phase II, pilot study to evaluate the efficacy and safety of apremilast involving 21 patients with PPP. The screening period was up to 4 weeks and treatment took place over 20 weeks per patient. No follow up period took place. No extension was done.

Recruitment period was 4 months; hence study duration from first patient in to last patient out was approximately 9 months. About 4-6 patients per center were recruited, assuming enrolment of both genders with distribution according to prevalence of condition.

Patient recruitment took place at 5 centers in Germany. The investigators had relevant expertise in diagnosing and treating PPP or were specialized in dermatology. Patients were enrolled until approximately 20 patients were included into the study. One drop-out was replaced during the recruitment phase.

Five visits per patient were performed including:

* Visit 1 at week -4 to -1 (screening)
* Visit 2 at week 0 (baseline)
* Visit 3 at week 4
* Visit 4 at week 12
* Visit 5 at week 20 (end of study)

After the end of study participation the investigator ensured that the patient received a suitable therapy appropriate to patient's condition.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients aged 18 years or more at screening visit.
* Patients with chronic PPP (disease history of at least 6 months of diagnosis), who were eligible for treatment with systemic therapy defined as having PPP inadequately controlled by topical treatment and/or phototherapy and/or previous systemic therapy
* Patients with chronic moderate to severe PPP defined as patients with a PPPASI ≥12 with or without concomitant plaque-type psoriasis
* Negative result of a urine pregnancy test taken at screening and at baseline for all women, except those who were surgically sterile or at least 1 year postmenopausal (i.e. at least 12 consecutive months with amenorrhea without other known or suspected medical cause)
* Willingness and capability of using a highly effective contraceptive measures from Screening visit until the end of at least one menstrual cycle (but not less than 28 days) following discontinuation of apremilast as defined below:

  * Female patient of childbearing potential (fertile, following menarche and until becoming post- menopausal unless permanently sterile) using a highly effective method of contraception OR female patients of non-childbearing potential (surgically sterilized [e.g. hysterectomy, bilateral salpingectomy and bilateral oophorectomy] or postmenopausal)
  * Male patient, and their female partner of childbearing potential, using a highly effective method of contraception
  * Adequate contraceptive method defined as:

    * A method with less than 1% failure rate (e.g. permanent sterilization, hormone implants, hormone injections, some intrauterine devices, or vasectomized partner) OR
    * The use of two methods of contraception (e.g. one barrier method [condom, diaphragm or cervical/vault caps] with spermicide and one hormonal contraceptive [e.g. combined oral contraceptives, patch, vaginal ring, injectables and implants])
* Patient was capable of understanding and giving written, voluntary informed consent before study screening.
* Willingness and capability of complying with all study procedure requirements, as per the Investigator's judgment (e.g. patient able to swallow the apremilast tablets, blood sampling).

Exclusion Criteria:

* General:

  * Pregnant or breast-feeding women
  * Current or history of psychiatric disease that would interfere with the ability to comply with the study protocol or give informed consent
  * Patients known to have had a substance abuse (drug or alcohol) problem within the previous 12 month
  * Individuals who were involved in the organization of the study
  * Patients who were in any way dependent on the investigator
  * Patients who were participating in a clinical study
  * Relatives, partner or staff of any clinical site personnel
* Disease-related:

  * Evidence of skin conditions (e.g. eczema) other than PPP/psoriasis that would interfere with evaluations of the effect of study medication on PPP or psoriasis.
  * Laboratory values from routine blood test taken within the 8 weeks prior to screening with any of the following:

    * Serum creatinine >1.4 x upper limit of normal (ULN) for age and gender
    * Estimated Glomerular Filtration Rate (eGFR) <30 mL/min/1.73m2 according to the Chronic Kidney Disease-Epidemiology Collaboration (CKD-EPI) equation
  * Pustular psoriasis lesions on the part of body other than hands or feet
  * Significant concurrent medical conditions at the time of screening, including:

    * Risk factors for renal toxicity (renal inflammation)
    * Severe hepatic dysfunction
    * Unstable angina pectoris
    * Uncompensated congestive heart failure
    * Severe pulmonary disease requiring hospitalization or supplemental oxygen therapy
    * Immunodeficiency disorders: primary or secondary
    * Known positive human immunodeficiency virus (HIV) test result, hepatitis B surface (HBS) antigen or hepatitis C virus (HCV) test result
    * Uncontrolled insulin-dependent diabetes mellitus
    * Cancer or history of cancer (except for resected cutaneous basal cell or squamous cell carcinoma) in the last 5 years
    * Open cutaneous ulcers
  * Any condition that, in the judgment of the investigator, might cause this study to be detrimental to the patient.
* Medication-related:

  * Ultraviolet B (UVB) therapy, topical steroids, topical calcineurin inhibitors, topical Vitamin A or D analog preparations, or anthralin within 14 days of baseline. Exceptions: low potency topical corticosteroids (class I and II, according to European classification for potency of topical corticosteroids) were allowed as therapy for the face, groin, axillae in accordance with the manufacturer's suggested usage dose
  * Psoralen plus ultraviolet A radiation (PUVA), ciclosporin, acitretin, alitretinoin, alefacept (Amevive®), anakinra (Kineret®), systemic corticosteroids, methotrexate, fumaric acids or any other systemic anti- psoriasis therapy within 28 days of baseline
  * Prior (within the last 2 years) or concomitant use of antipsoriatic biologic therapy with TNF-alpha blocker and/or ustekinumab and/or ixekizumab and/or secukinumab and/or brodalumab and/or guselkumab
  * Concomitant use of strong cytochrome P450 3A4 (CYP3A4) enzyme inductors (e.g. rifampicin, phenobarbital, carbamazepin, phenytoin and St. John's wort)
  * Use of an investigational drug within 4 weeks prior to baseline or 5 pharmacokinetic/pharmacodynamics half-lives (whichever is longer)
  * Prior treatment with apremilast/Otezla®
  * Receipt of any live (attenuated) vaccine within 28 days prior to baseline
  * Concomitant use of any other PDE4 inhibitor
  * Patients with hereditary problems of galactose intolerance, lapp lactase deficiency or glucose-galactose malabsorption
  * For patients with skin biopsy samples taken: patients with clinically relevant coagulation disorders or medication or known hypersensitivity against local anesthetics.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2018-11-29 (Actual); Primary Completion 2019-08-29 (Actual); Study Completion 2019-08-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kristian Reich, MD, PhD, Study Chair — Prof. Dr. Kristian Reich
Locations (5):
- Germany (5):
  - University Hospital Bonn, Bonn
  - Universitätsmedizin Göttingen / Georg-August-Universität Department for Dermatology, Venereology and Allergology, Göttingen
  - SCIderm GmbH, Harburg
  - Universitätsklinik Schleswig-Holstein, Campus Kiel, PSORIASIS-ZENTRUM KIEL, Klinik für Dermatologie, Venerologie und Allergologie, Kiel
  - Universitätsklinikum Münster Klinik für Hautkrankheiten, Münster

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Wilsmann-Theis D, Kromer C, Gerdes S, Linker C, Magnolo N, Sabat R, Reich K, Mossner R. A multicentre open-label study of apremilast in palmoplantar pustulosis (APLANTUS). J Eur Acad Dermatol Venereol. 2021 Oct;35(10):2045-2050. doi: 10.1111/jdv.17441. Epub 2021 Jun 24. PMID 34077577

RESULTS

PARTICIPANT FLOW:
Groups:
- Full Analysis Set (FAS): The full analysis set (FAS) consisted of all patients who received at least one dose of study drug.
  Apremilast was taken orally twice daily (except Day 1). During the first 5 days, the dosage was up-titrated. The initial dose on day 1 was 10 mg in the morning; this was increased to 10 mg in the morning and evening on day 2. The evening dose was further increased by 10 mg (to 20 mg) on day 3. On day 4, the morning dose was increased to 20 mg, so that 20 mg was taken twice daily, and on day 5 the evening dose was increased to 30 mg. From Day 6 onwards, patients received the 30 mg dose twice a day.
Period: Overall Study
Arm/Group | Full Analysis Set (FAS)
Started | 21
Completed | 20
Not Completed | 1
Not completed — Adverse Event | 1

BASELINE CHARACTERISTICS:
Arm/Group | Full Analysis Set (FAS)
Number analyzed (Participants) | 21
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.76 (9.26)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16
  Male | 5
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: White | 20
  Race: Other (Sinti) | 1
Highest educational status [Count of Participants; unit: Participants]
  University degree | 2
  Professional School | 5
  Secondary school leaving certificate | 14
Is the patient a smoker? [Count of Participants; unit: Participants]
  Non-smoker | 2
  Ex-smoker | 4
  Current smoker | 15
Current involvement of scalp [Count of Participants; unit: Participants]
  No | 20
  Yes | 1
Current involvement of nails [Count of Participants; unit: Participants]
  No | 11
  Yes | 9
  Unknown | 1
Psoriatic arthritis [Count of Participants; unit: Participants] — Three patients (14.3%) were previously diagnosed with psoriatic arthritis, although one of these diagnoses was not verified by a rheumatologist.
  Participants
    No | 18
    Yes | 3
Psoriasis erythrodermica [Count of Participants; unit: Participants]
  No | 21
  Yes | 0
Psoriasis inversa [Count of Participants; unit: Participants]
  No | 19
  Yes | 2
Psoriasis pustulosa generalisata [Count of Participants; unit: Participants]
  No | 21
  Yes | 0
Plaque Psoriasis [Count of Participants; unit: Participants]
  No | 15
  Yes | 6
Do you suffer from P. vulgaris? [Count of Participants; unit: Participants]
  No | 15
  Yes | 6
Age at initial diagnosis of PPP [Mean (Standard Deviation); unit: years] | 52.10 (13.58)
Number of involved Fingernails [Mean (Full Range); unit: nails] | 1.22 [0.0 to 5.0]
Number of involved Toenails [Mean (Full Range); unit: nails] | 3.33 [0.0 to 9.0]

OUTCOME MEASURES:

1. Primary Outcome: Palmoplantar Pustulosis Psoriasis Area and Severity Index (PPPASI) at Week 20 Compared With Baseline
Description: The PPPASI assess palms of hands and soles of feet for psoriasis involvement. The PPPASI score range from 0-72, with higher scores indicating more severe disease.
Time Frame: PPPASI Score at baseline and Week 20.
Measure: Median (Inter-Quartile Range); unit: PPPASI Score
Groups:
- Per Protocol Set (PPS): The per protocol set (PPS) consisted of all patients who received at least one dose of study drug who completed the study with no major protocol violations.
- Full Analysis Set - LOCF: The full analysis set (FAS) consisted of all patients who received at least one dose of study drug. Missing values were imputed by the Last Observation Carried Forward (LOCF) method.
Arm/Group | Full Analysis Set (FAS) | Per Protocol Set (PPS) | Full Analysis Set - LOCF
Number analyzed (Participants) | 21 | 20 | 21
PPPASI Score
  Visit 2 - Baseline | 16.50 [14.00 to 19.50] | 15.85 [13.95 to 19.85] | 16.50 [14.00 to 19.50]
  Visit 5 - End of Study - Week 20 | 7.65 [4.45 to 10.6] | 7.65 [4.45 to 10.60] | 8.10 [4.50 to 11.20]
Statistical Analysis 1: Comparison: Full Analysis Set (FAS) vs Per Protocol Set (PPS); Test type: Other; p < 0.0001, Wilcoxon (Mann-Whitney); Wilcoxon Signed-rank test

2. Secondary Outcome: Number of Participants With PPPASI 50 Response
Description: PPPASI 50 response defined as a 50% decrease in PPPASI from baseline.
Time Frame: At Visit 3 (Week 4), Visit 4 (Week 12) and Visit 5 (Week 20).
Measure: Count of Participants; unit: Participants
Arm/Group | Full Analysis Set (FAS) | Per Protocol Set (PPS)
Number analyzed (Participants) | 21 | 20
Participants
  Visit 3 - Week 4 | 7 | 7
  Visit 4 - Week 12 | 12 | 12
  Visit 5 - End of Study - Week 20 | 13 | 13

3. Secondary Outcome: Number of Participants With PPPASI 75 Response
Description: PPPASI 75 response defined as a 75% decrease in PPPASI from baseline.
Time Frame: At Visit 3 (Week 4), Visit 4 (Week 12) and Visit 5 (Week 20).
Measure: Count of Participants; unit: Participants
Arm/Group | Full Analysis Set (FAS) | Per Protocol Set (PPS)
Number analyzed (Participants) | 21 | 20
Participants
  Visit 3 - Week 4 | 2 | 2
  Visit 4 - Week 12 | 6 | 6
  Visit 5 - End of Study - Week 20 | 3 | 3

4. Secondary Outcome: Dermatology Life Quality Index (DLQI)
Description: The DLQI is a dermatology-specific quality of life instrument designed to assess the impact of a disease on the patient's daily life which is also validated for PPP. It is a 10-item questionnaire and can be used to assess 6 different aspects: symptoms and feelings, leisure, daily activities, work or school performance, personal relationship and treatment. The DLQI was calculated by summing the score of each question resulting in a maximum of 30 and a minimum of 0. The higher the score, the more quality of life was impaired.
  Meaning of DLQI scores:
  * 0 to 1 = No effect at all on patient's life
  * 2 to 5 = Small effect on patient's life
  * 6 to 10 = Moderate effect on patient's life
  * 11 to 20 = Very large effect on patient's life
  * 21 to 30 = Extremely large effect on patient's life
Time Frame: At Visit 2 (Baseline), Visit 4 (Week 12) and Visit 5 (Week 20).
Population: The number analyzed in one or more rows differs from the overall number of patients included in the FAS or PPS population as DLQI score was not available for all patients at all timepoints.
Measure: Median (Inter-Quartile Range); unit: DLQI Score
Arm/Group | Full Analysis Set (FAS) | Per Protocol Set (PPS)
Number analyzed (Participants) | 21 | 20
DLQI Score
  Visit 2 - Baseline: number analyzed (Participants) | 20 | 19
  Visit 2 - Baseline | 8.50 [5.00 to 15.50] | 8.00 [5.00 to 16.00]
  Visit 4 - Week 12: number analyzed (Participants) | 20 | 20
  Visit 4 - Week 12 | 2.50 [1.00 to 10.50] | 2.50 [1.00 to 10.50]
  Visit 5 - End of Study - Week 20: number analyzed (Participants) | 19 | 19
  Visit 5 - End of Study - Week 20 | 2.00 [1.00 to 13.00] | 2.00 [1.00 to 13.00]

5. Other Pre Specified Outcome: Hand and Feet Physician Global Assessment (H&F PGA)
Description: The H&F PGA describes the severity of psoriasis on the hands and/or feet using five categories ranging from 0 (clear) to 4 (severe).
Time Frame: At Visit 2 (Baseline), Visit 3 (Week 4) , Visit 4 (Week 12) and Visit 5 (Week 20).
Population: In the FAS 20 participants were analyzed in all visits, except at Visit 2 (n=21).
Measure: Count of Participants; unit: Participants
Arm/Group | Full Analysis Set (FAS) | Per Protocol Set (PPS)
Number analyzed (Participants) | 21 | 20
Participants
  Visit 2 - Baseline: 0 clear | 0 | 0
  Visit 2 - Baseline: 1 almost clear | 0 | 0
  Visit 2 - Baseline: 2 mild | 2 | 2
  Visit 2 - Baseline: 3 moderate | 19 | 18
  Visit 2 - Baseline: 4 severe | 0 | 0
  Visit 3 - Week 4: number analyzed (Participants) | 20 | 20
  Visit 3 - Week 4: 0 clear | 0 | 0
  Visit 3 - Week 4: 1 almost clear | 1 | 1
  Visit 3 - Week 4: 2 mild | 10 | 10
  Visit 3 - Week 4: 3 moderate | 9 | 9
  Visit 3 - Week 4: 4 severe | 0 | 0
  Visit 4 - Week 12: number analyzed (Participants) | 20 | 20
  Visit 4 - Week 12: 0 clear | 0 | 0
  Visit 4 - Week 12: 1 almost clear | 3 | 3
  Visit 4 - Week 12: 2 mild | 9 | 9
  Visit 4 - Week 12: 3 moderate | 8 | 8
  Visit 4 - Week 12: 4 severe | 0 | 0
  Visit 5 - End of Study - Week 20: number analyzed (Participants) | 20 | 20
  Visit 5 - End of Study - Week 20: 0 clear | 1 | 1
  Visit 5 - End of Study - Week 20: 1 almost clear | 1 | 1
  Visit 5 - End of Study - Week 20: 2 mild | 10 | 10
  Visit 5 - End of Study - Week 20: 3 moderate | 8 | 8
  Visit 5 - End of Study - Week 20: 4 severe | 0 | 0

6. Other Pre Specified Outcome: Pustules Count Percent Change From Baseline
Description: Percentage change from baseline in Pustules count after 20 weeks of treatment with Apremilast
Time Frame: At Visit 2 (Baseline) and Visit 5 (End of Study - Week 20)
Measure: Median (Inter-Quartile Range); unit: Percent change
Arm/Group | Full Analysis Set - LOCF | Per Protocol Set (PPS)
Number analyzed (Participants) | 21 | 20
Percent change | -76.3 [-100 to -53.4] | -79.82 [-100 to -57.33]
Statistical Analysis 1: Comparison: Full Analysis Set - LOCF; Test type: Other; p < 0.001, Wilcoxon Signed-rank test

7. Other Pre Specified Outcome: Number of Participants With Pustules Count 50 and 75 Response
Description: Patients experiencing a 50% and 75% decrease in Pustules count from baseline
Time Frame: At Visit 3 (Week 4), Visit 4 (Week 12) and Visit 5 (End of Study-Week 20).
Measure: Count of Participants; unit: Participants
Arm/Group | Full Analysis Set (FAS) | Per Protocol Set (PPS)
Number analyzed (Participants) | 21 | 20
Participants
  Pustules count 50: Visit 3 - Week 4 | 13 | 14
  Pustules count 50: Visit 4 - Week 12 | 18 | 17
  Pustules count 50: Visit 5-End of Study- Week 20 | 16 | 16
  Pustules count 75: Visit 3 - Week 4 | 8 | 9
  Pustules count 75: Visit 4 - Week 12 | 14 | 14
  Pustules count 75: Visit 5-End of Study- Week 20 | 12 | 12

8. Other Pre Specified Outcome: Visual Analogue Scale (VAS) Discomfort/Pain
Description: VAS was used to assess discomfort/pain. The patient was asked to place a vertical stroke on a 100 mm VAS on which the left-hand boundary represented no discomfort/pain (at 0 mm), and the right-hand boundary (at 100 mm) represented discomfort/pain as severe as can be imagined. The distance from the mark to the left-hand boundary was recorded, with higher values indicating more discomfort/pain (worse conditions).
Time Frame: At Visit 2 (Baseline), Visit 3 (Week 4), Visit 4 (Week 12) and Visit 5 (End of Study - Week 20).
Measure: Median (Inter-Quartile Range); unit: Units on a scale
Arm/Group | Full Analysis Set (FAS) | Per Protocol Set (PPS)
Number analyzed (Participants) | 21 | 20
Units on a scale
  Visit 2 - Baseline | 44.0 [11.0 to 67.0] | 37.5 [9.0 to 61.0]
  Visit 3 - Week 4 | 4.0 [0.0 to 19.0] | 3.0 [0.0 to 19.0]
  Visit 4 - Week 12 | 2.0 [0.0 to 27.0] | 1.5 [0.0 to 21.0]
  Visit 5 - End of Study - Week 20 | 9.0 [3.0 to 61.0] | 7.5 [2.5 to 29.5]

9. Other Pre Specified Outcome: Visual Analogue Scale (VAS) Pruritus/Itch
Description: VAS was used to assess pruritus/itch. The patient was asked to place a vertical stroke on a 100 mm VAS on which the left-hand boundary (at 0 mm) represented no pruritus/itch, and the right-hand boundary (at 100 mm) represented pruritus/itch as severe as can be imagined. The distance from the mark to the left-hand boundary was recorded, with higher values indicating more pruritus/itch (worse outcomes).
Time Frame: At Visit 2 (Baseline), Visit 3 (Week 4), Visit 4 (Week 12) and Visit 5 (End of Study - Week 20).
Measure: Median (Inter-Quartile Range); unit: Units on a scale
Arm/Group | Full Analysis Set (FAS) | Per Protocol Set (PPS)
Number analyzed (Participants) | 21 | 20
Units on a scale
  Visit 2 - Baseline | 31.0 [16.0 to 55.0] | 29.5 [12.5 to 49.0]
  Visit 3 - Week 4 | 2.0 [2.0 to 48.0] | 11.0 [2.0 to 39.75]
  Visit 4 - Week 12 | 25.0 [4.0 to 44.0] | 24.0 [3.5 to 37.25]
  Visit 5 - End of Study - Week 20 | 12.0 [6.0 to 49.0] | 11.5 [5.25 to 30.25]

10. Other Pre Specified Outcome: Psoriasis Area and Severity Index (PASI)
Description: The PASI is a measure of psoriatic disease severity taking into account qualitative lesion characteristics (erythema, thickness, and scaling) and degree of skin surface area involvement on defined anatomical regions. PASI scores range from 0 to 72, with higher scores reflecting greater disease severity. Erythema, thickness, and scaling are scored on a scale of 0 (none) to 4 (very severe) on 4 anatomic regions of the body: head, trunk, upper limbs, and lower limbs. Degree of involvement on each of the 4 anatomic regions is scored on a scale of 0 (no involvement) to 6 (90% to 100% involvement). The total qualitative score (sum of erythema, thickness, and scaling scores) is multiplied by the degree of involvement for each anatomic region and then multiplied by a constant. These values for each anatomic region are summed to yield the PASI score.
Time Frame: At Visit 2 (Baseline), Visit 3 (Week 4), Visit 4 (Week 12) and Visit 5 (End of Study - Week 20).
Population: PASI score was available only for 6 patients included in the PPS population at all assessment times.
Measure: Median (Inter-Quartile Range); unit: PASI Score
Arm/Group | Per Protocol Set (PPS)
Number analyzed (Participants) | 6
PASI Score
  Visit 2 - Baseline | 3.85 [1.93 to 5.18]
  Visit 3 - Week 4 | 2.27 [0.3 to 3.65]
  Visit 4 - Week 12 | 0.5 [0.0 to 2.35]
  Visit 5-End of Study-Week 20 | 0.95 [0.0 to 2.28]

11. Other Pre Specified Outcome: Dynamic H&F PGA
Description: The dynamic H&F PGA describes the global improvement compared with baseline. It relies on the physician's memory of the baseline severity to evaluate the level of alteration. The categories vary between 0 (cleared) and 6 (worse).
Time Frame: At Visit 3 (Week 4), Visit 4 (Week 12) and Visit 5 (End of Study - Week 20).
Measure: Count of Participants; unit: Participants
Arm/Group | Per Protocol Set (PPS)
Number analyzed (Participants) | 20
Participants
  Visit 3 - Week 4: 0 cleared | 0
  Visit 3 - Week 4: 1 excellent | 2
  Visit 3 - Week 4: 2 good | 4
  Visit 3 - Week 4: 3 slight | 3
  Visit 3 - Week 4: 4 unchanged | 4
  Visit 3 - Week 4: 5 fair | 7
  Visit 3 - Week 4: 6 worse | 0
  Visit 4 - Week 12: 0 cleared | 0
  Visit 4 - Week 12: 1 excellent | 5
  Visit 4 - Week 12: 2 good | 5
  Visit 4 - Week 12: 3 slight | 2
  Visit 4 - Week 12: 4 unchanged | 2
  Visit 4 - Week 12: 5 fair | 6
  Visit 4 - Week 12: 6 worse | 0
  Visit 5 - End of Study - Week 20: 0 cleared | 0
  Visit 5 - End of Study - Week 20: 1 excellent | 5
  Visit 5 - End of Study - Week 20: 2 good | 7
  Visit 5 - End of Study - Week 20: 3 slight | 2
  Visit 5 - End of Study - Week 20: 4 unchanged | 2
  Visit 5 - End of Study - Week 20: 5 fair | 4
  Visit 5 - End of Study - Week 20: 6 worse | 0

ADVERSE EVENTS:
Time Frame: All AEs were monitored/assessed from baseline (Visit 2, onset of treatment) until the patient's last study visit (i.e., up to 20 weeks). All SAEs were monitored/assessed upon ICF signature (Visit 1) until 30 days after the patient had stopped study participation (i.e., up to 24 weeks plus 30 days).
Description: The date of onset, intensity, relationship of the AE to study drug, action(s) taken, seriousness, time course, duration and outcome were recorded.
Arm/Group | Full Analysis Set (FAS)
All-Cause Mortality (participants affected / at risk) | 0/21
Serious Adverse Events (participants affected / at risk) | 0/21
Other Adverse Events (participants affected / at risk) | 19/21
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Full Analysis Set (FAS) (N=21)
Arthropod bite (Injury, poisoning and procedural complications) | 3 (3)
Post procedural swelling (Injury, poisoning and procedural complications) | 1 (1)
Ligament sprain (Injury, poisoning and procedural complications) | 1 (1) — No treatment-emergent
Artificial crown procedure (Surgical and medical procedures) | 1 (1)
Endodontic procedure (Surgical and medical procedures) | 1 (1)
Tachycardia (Cardiac disorders) | 1 (1)
Nasal dryness (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Headache (Nervous system disorders) | 5 (7)
Nerve compression (Nervous system disorders) | 1 (1)
Tension headache (Nervous system disorders) | 1 (1) — No treatment-emergent
Chest discomfort (General disorders) | 1 (1)
Anxiety disorder (Psychiatric disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 6 (6)
Diarrhoea (Gastrointestinal disorders) | 5 (6)
Abdominal pain (Gastrointestinal disorders) | 2 (2)
Abdominal pain upper (Gastrointestinal disorders) | 2 (2)
Epulis (Gastrointestinal disorders) | 1 (1)
Flatulence (Gastrointestinal disorders) | 1 (1)
Gastritis (Gastrointestinal disorders) | 1 (1)
Toothache (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
Actinic keratosis (Skin and subcutaneous tissue disorders) | 1 (1)
Dermatitis (Skin and subcutaneous tissue disorders) | 1 (1)
Eczema (Skin and subcutaneous tissue disorders) | 1 (1)
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Exostosis (Musculoskeletal and connective tissue disorders) | 1 (1)
Intervertebral disc disorder (Musculoskeletal and connective tissue disorders) | 1 (1)
Limb discomfort (Musculoskeletal and connective tissue disorders) | 1 (1)
Tendonitis (Musculoskeletal and connective tissue disorders) | 1 (1)
Nasopharyngitis (Infections and infestations) | 5 (6) — One event of nasopharyngitis was no treatment-emergent
Cystitis (Infections and infestations) | 1 (1)
Gastrointestinal infection (Infections and infestations) | 1 (1)
Influenza (Infections and infestations) | 1 (1)
Respiratory tract infection (Infections and infestations) | 1 (1)
Sinusitis (Infections and infestations) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1) — No treatment-emergent

LIMITATIONS AND CAVEATS:
The interpretation of APLANTUS study is limited by the short-term 20-week treatment period and the size of the population.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2018-06-07): https://cdn.clinicaltrials.gov/large-docs/97/NCT04572997/Prot_000.pdf
  • Statistical Analysis Plan (2019-06-20): https://cdn.clinicaltrials.gov/large-docs/97/NCT04572997/SAP_001.pdf